CLINICAL TRIAL: NCT04467086
Title: Propranolol as an Anxiolytic to Reduce the Use of Sedatives From Critically-ill Adults Receiving Mechanical Ventilation: An Open-label Randomized Controlled Trial (PROACTIVE)
Brief Title: Propranolol as an Anxiolytic to Reduce the Use of Sedatives From Critically-ill Adults Receiving Mechanical Ventilation
Acronym: PROACTIVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Hamilton Health Sciences Corporation (Other); The Ottawa Hospital (Other); McMaster University (Other); Sinai Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 776228483
Record Dates: First submitted 2020-06-30; First posted 2020-07-10 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Mechanical Ventilation; Sedation; Critical Illness; COVID
Keywords: randomized clinical trial; phase III; propranolol; sedative use; sedative sparing; sedative shortages; critical care; cost savings
MeSH Terms: conditions — Critical Illness | interventions — Propranolol

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial with 1:1 allocation (intervention and control group)
Who Masked: Participant
Masking Description: Participants will be masked to intervention versus control group allocation. Care providers (including investigators) cannot be masked due to the need to titrate propranolol and sedative doses according to patient condition in the intervention arm. Similarly, outcomes assessors will be recording the daily and total doses of propranolol received by each participant, and thus cannot be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Arm - Usual Care (No Intervention): Participants in the control group will receive usual intravenous sedation according to practices already in place at each participating site. The choice of agent, route of delivery, method of monitoring, and target levels of sedation will be determined by the treating team; however, we will recommend best practice clinical guidelines be followed. Current guidelines recommend "analgesia first" sedation titrated to relief of pain and dyspnea and sedative infusions if need for anxiety or agitation titrated to a prescribed level of sedation using a validated sedation scale. Patients may receive adjunct sedative/analgesic medications (e.g., enteral benzodiazepines) but propranolol use in the control group will be considered a protocol violation.
- Intervention Arm - Propranolol hydrochloride (Experimental): Participants in the control arm will received sedation as described for the control arm, but with the addition of propranolol hydrochloride (titrated up as described under "Intervention Description") and a corresponding reduction in sedatives as appropriate and described under "Intervention Description".
  Interventions: Drug: Propranolol Hydrochloride

INTERVENTIONS:
Drug: Propranolol Hydrochloride — Propranolol enterally at a starting dose of 20mg every 6h for 2-4 doses, and then re-assessed for upwards titration every 24 hours (+/- 6 hours) at 10mg dose increases depending on clinical response. Maximum dose of 60mg every 6h. Titration decision to be made by clinical team at daily rounds.
  Daily titration will be guided by hemodynamic markers indicative of the expected sympatholysis from propranolol. Upward titration of propranolol should coincide with a downward titration in sedatives until a minimum level of sedative infusion is reached (propofol <0.5mg/kg/h or midazolam <1.0mg/h). Nurses will be instructed at each assessment to determine if sedative targets can be achieved with lower doses of sedatives. Daily upward titration of propranolol will be recommended if none of these conditions are met: (1)HR<70 beats/min, (2) Mean Arterial Pressure <70 mmHg or (3) norepinephrine or equivalent vasopressor dose increase to >0.15 mcg/kg/min.
  Other Names: Teva-propranolol
  Arms: Intervention Arm - Propranolol hydrochloride

SUMMARY:
The COVID-19 pandemic has led to shortages of intravenous sedatives due to increased ICU patient admissions and greater use of mechanical ventilation. A shortage of sedatives is as concerning as a shortage of mechanical ventilators since critically ill patients require sedation for comfort and to tolerate mechanical ventilation. Anti-adrenergic medications are increasingly recognized for their role in sedation of critically ill patients. Propranolol is a plentiful and inexpensive, non-selective beta-adrenergic blocker with good penetration of the blood-brain barrier, which can reduce agitation and arousal. The study team published a single-centre retrospective study of 64 mechanically-ventilated patients which found the initiation of propranolol was associated with an 86% reduction in propofol dose and a roughly 50% reduction in midazolam dose while maintaining the same level of sedation. Propranolol has the potential to mitigate the threat posed by worldwide sedative shortages and improve critical care management of patients who require mechanical ventilation.

This study seeks to evaluate whether the addition of propranolol to a standard sedation regimen reduces the dose of sedative needed in critically ill patients requiring mechanical ventilation. This study is an open-label randomized controlled trial, single-blinded with 1:1 allocation. Both arms will receive sedation according to usual intensive care unit practice with a sedative agent. The intervention arm will additionally receive enteral propranolol 20-60mg q6h titrated up over 24-48h until intravenous sedative doses have fallen to a minimal level (propofol <0.5mg/kg/h or midazolam <0.5mg/h) or the maximum dose of propranolol is reached. Intravenous sedative doses will be titrated downwards in response to sympatholysis produced by the propranolol, as evidenced by a decreasing heart rate or blood pressure. The control arm will receive sedation without the addition or propranolol.

The primary outcome will be the change in primary sedative dose from baseline to Day 3 of enrollment. Analysis of the primary outcome will be a difference in differences; the change in sedative dose from baseline to Day 3 in the intervention group versus the same change in the control group. The Mann-Whitney U test will be used as a nonparametric test of independent samples for this outcome.

DETAILED DESCRIPTION:
Background and Rationale:

Critically ill patients often require sedation for comfort and to tolerate mechanical ventilation. There are internationally accepted guidelines for sedation of critically ill patients, and dexmedetomidine and propofol are recommended as sedative agents over alternatives, such as benzodiazepines. There is now a worrying shortage of propofol in Canada, the European Union, and parts of the US. The supply of dexmedetomidine, an expensive alternative to propofol, is now considered to be at risk. It is unsuitable as monotherapy for deep sedation, and most hospitals in Canada limit use to 48h, due to high costs. This therefore makes it inadequate for COVID-19 treatment. Other sedative agents for mechanical ventilation include benzodiazepines (e.g. midazolam), but these are associated with higher mortality from sepsis, higher incidence of delirium, and longer length of stay in the ICU. That notwithstanding, midazolam is also currently in short supply. Shortages of sedative medications will be as impactful on critical care practice as shortages of mechanical ventilators; propofol, midazolam, and dexmedetomidine were all listed on March 31, 2020 as "Tier 3 Shortages" by Health Canada - having "the greatest potential impact on Canada's drug supply and health care system….based on low availability of alternative supplies, ingredients or therapies."

In critically-ill patients, the sympathetic nervous system can become hyperactive, producing neurotransmitters such as norepinephrine (NE) to increase blood pressure and heart rate. In the brain, a pontine nucleus called the locus ceruleus (LC) provides the majority of brain NE. LC adrenergic input to the medial septal area and medial preoptic area of the forebrain mediates arousal.

Sympatholytics have previously been prescribed to manage agitation in critical illness. Dexmedetomidine is one such example, an intravenous alpha-2 agonist, which readily penetrates the central nervous system. It has an anti-noradrenergic effect in the locus ceruleus, consequently increasing inhibitory GABA neuron activity in the forebrain. Clonidine, is an oral and intravenous agent that is highly lipid soluble, with good penetration of the Central Nervous System, has been well studied in the ICU environment. However a recent meta-analysis showed clonidine use did not reduce length of stay or length of ventilation for critically ill patients, and only led to a small reduction in the use of opioids. Propranolol is a non-selective beta-adrenergic antagonist, approved for treating hypertension, angina, arrhythmias, migraines and pheochromocytoma in Canada. It has also been used off label to treat anxiety disorders such as Post-Traumatic Stress Disorder. It is a lipophilic molecule, crosses the blood brain barrier, and can block the locus ceruleus' ability to activate the forebrain, similar to alpha 2 agonists. In rat models, propranolol delays arousal from a state of anaesthesia.

An extensive search of PubMed and Web of Science did not reveal published trials of propranolol as a sedative agent in critical illness or mechanical ventilation. However, propranolol was shown to significantly reduce agitation in a randomized controlled trial in patients with traumatic brain injury. Observational studies in traumatic brain injury have shown that propranolol use is associated with a shorter length of hospital and ICU stay, and possibly a lower mortality risk, without reports of significant side effects. A meta-analysis of 10 randomized controlled trials in severely burned patients found propranolol reduced hospital length of stay. Other studies have shown that propranolol may have beneficial effects on catabolism in critical illness, and improve cardiac function and survival in animal models of cardiac resuscitation. This study team published a single centre retrospective study of 64 mechanically-ventilated patients which found that the initiation of propranolol was associated with an 86% reduction in propofol dose, and an approximately 50% reduction in midazolam dose, while maintaining the desired sedation target.

If propranolol reduces sedative doses required by mechanically ventilated patients (either with or without COVID illness) to the degree seen in this team's retrospective study, this would effectively reduce usage of sedatives two- to seven-fold. The cost of the average daily dose of propranolol used in the retrospective study (~120mg) would be $0.27 (pharmacy cost at The Ottawa Hospital), and propranolol is in abundant supply in Canada and around the world.

Based on this data, propranolol may enable critical care providers to sedate mechanically ventilated patients using their usual approaches except with substantially lower doses of sedatives. This would not only extend the use of currently limited supply of sedatives, it would significantly reduce medication costs in critical care units in Canada and worldwide.

Trial Objective:

Does the addition of propranolol to a standard sedation regimen reduce the dose of sedative needed in critically ill patients requiring mechanical ventilation?

Study Design:

Open-label, Randomized Controlled Trial (RCT), 1:1 allocation

Patient Population:

Participants are adult patients admitted to an intensive care unit who are anticipated to require mechanical ventilation >48h, who are requiring intravenous sedatives to achieve a sedation goal that is anticipated to be stable for >48h.

Intervention:

Patients randomized to the intervention arm will receive propranolol enterally at a starting dose of 20mg every 6 hours for two to four doses, and then re-assessed for upwards titration every 24 hours (+/- 6 hours) at 10mg dose increases depending on clinical response. The maximum dose to be used in the intervention group is 60mg every 6 hours. The decision to titrate propanolol will be made daily at rounds; this is why participants will receive 2-4 doses at 20mg (to accommodate for time from enrollment to rounds the next day) and titration will occur every 24 hours +/- 6 hours (to accommodate rounds timing). Titration timing is based on clinical rounds so that the decision to titrate can be made by the clinical team in a way that aligns with their clinical workflows and reflects actual clinical practice in the ICU.

Daily dose titration will be guided by hemodynamic markers indicative of the expected sympatholysis from propranolol. Upward titration of propranolol should coincide with a downward titration in sedatives until a minimum level of sedative infusion is reached (propofol <0.5mg/kg/h or midazolam <0.5mg/h). For each participant, the intervention will be administered from enrollment until approximately 48h after the patient is liberated from the mechanical ventilator, and the study will continue until death, ICU discharge, or 30 days after enrollment, whichever is first. Enrollment can begin as early as 24h after the start of a sedative infusion in the ICU.

Primary Outcome and Sample Size:

The primary outcome will be a comparison of the change in primary sedative dose from baseline to Day #3 of the study in the intervention group compared with the same change in the control group- the difference in differences. Given the global need for a substantial reduction in sedative consumption for mechanically ventilated patients, we will assume that a 70% reduction in sedative dose would be clinically meaningful, which corresponds to the difference between the sedative infusion doses required for study eligibility (ie. propofol >1.5 mg/kg/h) and the minimum doses below which propranolol would no longer be increased (ie. propofol <0.5 mg/kg/h). Since we do not have (or know of) any data with which to estimate the standard deviation of the change in sedative use, we base our sample size calculation on the Cohen's d statistic (also known as the standardized effect size). The standardized effect size is computed as the magnitude of the difference between groups divided by the pooled standard deviation of the response measure (in our case, the change in sedative dose from baseline to day 3). By widespread consensus, standardized effect sizes of 0.2, 0.5, and 0.8 are respectively considered to be small, moderate, and large effect sizes. Given we would need to see at least a moderately large change in sedative use (decrease of 70%) to effect a substantial improvement in the overall sedative supply, we choose to power our trial to detect a standardized effect of 0.5. In order to have 80% power to detect such a minimal clinically important difference, we require a total of 32 participants in each study arm. in a 1:1 randomized controlled trial. Allowing a 10% dropout rate (a previous study of sedation strategies at these sites reported a dropout rate of 3%30), we will aim to enroll 72 patients (36 control; 36 intervention).

Statistical Analysis:

The primary outcome will be analyzed as a difference in differences- the change in sedative dose from baseline to Day #3 (defined as the 24h period starting 60h after enrollment) in the intervention group vs the same change in the control group. The Mann-Whitney U test will be used as a nonparametric test of independent samples for this outcome, as well as the secondary outcomes that relate to sedative dosing on Day #3 compared to baseline. For secondary outcomes, groups will be compared using unpaired statistical tests- Chi-square for proportions, and unpaired t-tests or Mann-Whitney tests as appropriate for parametric and non-parametric data. The effect of age, sex and gender, and pre-ICU beta-blocker prescription will be analyzed as planned subgroup analyses.

Ethical Considerations:

A No Objection Letter from Health Canada and Research Ethics Board approval have been obtained to conduct this clinical trial. An established data safety monitoring committee (DSMC) will evaluate adverse events. Two interim safety analyses will be conducted by the DSMC and the study will be terminated if the DSMC determines the risk of adverse events, based on the rate of adverse events reported in this clinical trial to the committee, outweighs the potential benefits. Informed consent will be obtained from each participant or their legal substitute decision maker.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted to an intensive care unit requiring mechanical ventilation and anticipated to require mechanical ventilation >48h
* Patient has a sedation target (e.g. using the Richmond Agitation Sedation Scale or Sedation Agitation Scale) that is anticipated to be stable >48h
* Minimum sedative infusion doses (any one of):

  * Propofol >/=1.5 mg/kg/h >24h
  * Midazolam >/=3.0 mg/h >24h

Exclusion Criteria:

* Sedation for paralysis
* Use of neuromuscular blocking agents (patients may be eligible once these are discontinued)
* Asthma or known reactive airways disease
* 1st, 2nd or 3rd-degree heart block (with no permanent pacemaker) at the time of screening
* Known history of congestive heart failure with ejection fraction <20%
* HR<60 bpm at baseline
* Hypotension requiring vasopressor support above the following levels

  * Norepinephrine dose >0.15mcg/kg/min or equivalent (>0.15mcg/kg/min epinephrine; >22.5 mcg/kg/min dopamine; >0.06 U/min vasopressin)
  * Phenylephrine >2.0 mcg/kg/min
  * Receiving 3 or more vasopressors, regardless of dose
* Pregnancy or lactation
* Allergy to propranolol
* Patients for whom an enteral route of drug administration is not available
* Patients who are on digoxin, diltiazem, or verapamil
* Patients on chronic betablockers are eligible for enrolment. Patients allocated to the intervention arm will have their betablocker replaced with propranolol. Once propranolol is discontinued, the treating team may resume their usual betablocker. Control patients may continue their usual betablocker (unless it is propranolol) at the treating team's discretion.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Primary sedative dose change | 24 hours prior to enrollment to Day 3 of the study (60-84hrs after enrollment)
  Change from baseline in total daily dose of primary sedative on Day 3

SECONDARY OUTCOMES:
Sedation scores | Daily upon enrollment until study completion (discharge from ICU, 28 days, or death - whichever is first)
  Proportion of measured sedation scores within target range (to be defined a priori by treating team): Richmond Agitation-Sedation Scale and/or the Sedation-Agitation Scale
Primary sedative dose | Day 3 of study (60-84hrs after enrollment)
  Proportion of participants whose sedative dose on day 3 are below a minimum level (propofol <0.5mg/kg/h or midazolam <1.9mg/h)
Total sedative daily dose change | 24 hours prior to enrollment to Day 3 of the study (60-84hrs after enrollment)
  Change from baseline in total daily dose of all sedatives (in mg of midazolam equivalents) on Day 3
Total opioid daily dose change | 24 hours prior to enrollment to Day 3 of the study (60-84hrs after enrollment)
  Change from baseline in total daily dose of all opioids (in mcg of fentanyl equivalents) on Day 3
Adverse event - bradycardia | Daily from study enrollment until study completion (discharge from ICU, 28 days, or death - whichever is first)
  Incidence of bradycardia (HR <50 or requiring intervention)
Adverse event - hypotension | Daily from study enrollment until study completion (discharge from ICU, 28 days, or death - whichever is first)
  Incidence of hypotension (MAP <60 requiring new vasopressor agents or an increase of >0.1 mcg/kg/min of norepinephrine or epinephrine persisting more than 2h after reducing sedative doses)
Adverse event - bronchospasm | Daily from study enrollment until study completion (discharge from ICU, 28 days, or death - whichever is first)
  Incidence of clinically-important bronchospasm requiring a change in mechanical ventilation settings
Adverse event - ECG conduction delays | Daily from study enrollment until study completion (discharge from ICU, 28 days, or death - whichever is first)
  Incidence of new ECG conduction delays

OTHER OUTCOMES:
Duration of propranolol use | Daily from enrollment to study withdrawal/completion (last day of propranolol dose given; discharge from ICU, 28 days, or death - whichever is first)
  Total number of days of propranolol use
Propranolol dose | Day 3 of study (60-84hrs after enrollment)
  Mean propranolol dose on day 3
Ventilator-free days | Day 1 of admission to the intensive care unit until 30 days, discharge from intensive care, or death (whichever is first)
  Mean number of ventilator-free days in first 30 days of hospital intensive care unit admission
Delirium-free days | Day 1 of admission to the intensive care unit until 30 days, discharge from intensive care, or death (whichever is first)
  Mean number of delirium-free days in first 30 days of hospital intensive care unit admission, measured using the Intensive Care Delirium Screening Checklist
Hospital Length of Stay | Day 1 of hospital admission until hospital discharge date or date of death (whichever is first)
  Mean length of stay in hospital
Intensive Care Unit Length of Stay | Day 1 of intensive care unit admission until discharge date from intensive care unit or date of death (whichever is first)
  Mean length of stay in the intensive care unit
Hospital Mortality | Upon study completion (after all 108 participants have completed the study, estimated at 6 months) and after 50 patients have been enrolled (estimated at 3 months)
  Mortality rate among participants while in hospital
Direct Costs | Upon study completion (after all 108 participants have completed the study, estimated at 6 months)
  Mean cost of sedative medication used in the intensive care unit among the intervention and control arms

CONTACTS AND LOCATIONS:
Overall Officials: James Downar, MDCM, Principal Investigator — Ottawa Hospital Research Institute
Locations (2):
- Canada (2):
  - Hamilton Health Sciences Centre - Hamilton General Hospital, Hamilton, Ontario
  - The Ottawa Hospital, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bergeron N, Dubois MJ, Dumont M, Dial S, Skrobik Y. Intensive Care Delirium Screening Checklist: evaluation of a new screening tool. Intensive Care Med. 2001 May;27(5):859-64. doi: 10.1007/s001340100909. PMID 11430542
- [Background] Sessler CN, Gosnell MS, Grap MJ, Brophy GM, O'Neal PV, Keane KA, Tesoro EP, Elswick RK. The Richmond Agitation-Sedation Scale: validity and reliability in adult intensive care unit patients. Am J Respir Crit Care Med. 2002 Nov 15;166(10):1338-44. doi: 10.1164/rccm.2107138. PMID 12421743
- [Background] Riker RR, Picard JT, Fraser GL. Prospective evaluation of the Sedation-Agitation Scale for adult critically ill patients. Crit Care Med. 1999 Jul;27(7):1325-9. doi: 10.1097/00003246-199907000-00022. PMID 10446827
- [Derived] Downar J, Lapenskie J, Kanji S, Watpool I, Haines J, Saeed U, Porteous R, Polskaia N, Burry L, Himed S, Anderson K, Fox-Robichaud A. Propranolol As an Anxiolytic to Reduce the Use of Sedatives for Critically Ill Adults Receiving Mechanical Ventilation (PROACTIVE): An Open-Label Randomized Controlled Trial. Crit Care Med. 2025 Feb 1;53(2):e257-e268. doi: 10.1097/CCM.0000000000006534. Epub 2025 Feb 21. PMID 39982178
- [Derived] Bertolini F, Robertson L, Bisson JI, Meader N, Churchill R, Ostuzzi G, Stein DJ, Williams T, Barbui C. Early pharmacological interventions for prevention of post-traumatic stress disorder (PTSD) in individuals experiencing acute traumatic stress symptoms. Cochrane Database Syst Rev. 2024 May 20;5(5):CD013613. doi: 10.1002/14651858.CD013613.pub2. PMID 38767196